CLINICAL TRIAL: NCT04217538
Title: Observational Study of a Cohort of Patients With Hereditary Epidermolysis Bullosa That Come for Their Annual/Biannual Check up at This Medical Rare Disease Reference Centers (MRDRC) of This Disease in France and Belgium
Brief Title: Observational Study of a Cohort of Patients With Hereditary Epidermolysis Bullosa
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 19-ODONTO-01
Record Dates: First submitted 2019-12-31; First posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EBH
  Interventions: Other: clinical exam

INTERVENTIONS:
Other: clinical exam — clinical oral examination

SUMMARY:
Hereditary Epidermolysis Bullosa (EBH) are rare dermatologic diseases characterized by cutaneous and mucosa fragility. Oral manifestations of few small cohort have been published. The main objective of this multicentric cohort study first in Europe was to report the oral status of these patients that were consulted in the MRDRC of this disease in Nice (France), Toulouse (France) and Louvain (Belgium). Then a correlation between the oral characteristics and the EBH type will be made, in order to facilitate the management of patient care and the prevention program that can be established to improve their oral health.

ELIGIBILITY:
Inclusion Criteria:

* patient with EBH
* patient consent for examination and use the clinical data for publication purpose

Exclusion Criteria:

-

Ages: 7 Months to 78 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients with EBH are recruted from the 2 MRDRC of the disease in France and the one of Belgium, the dental visit was/is organized for each visit/follow up of the patient in the center (annual or bianual visit)
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Dental structural abnormalities and/or caries | 1 day
  number of defect /dental caries dor each toth

SECONDARY OUTCOMES:
gingival biotype | 1 day
  clinical observation of gingiva (thin or thick)
gingival status | 1 day
  observation and classification of the gingiva (healthy, inflammed or hyperplastic)
plaque and gingival index | 1 day
  registration of plaque and gingival index according to the Loë and Silness method
oral lesion | 1 day
  number and localisation of the blister/scars/flanges scars on a sketch of a mouth

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Nice Hospital, Nice
  - Toulouse University, Toucy